CLINICAL TRIAL: NCT05260827
Title: The Effects of Heated Tobacco Products Use on Lung Function and Volatile Organic Compounds in Exhaled Air
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Magnus Lundbäck, PI, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Karolinska Institutet 2
Record Dates: First submitted 2021-10-08; First posted 2022-03-02 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Lung Inflammation
Keywords: lung function; volatile organic compounds; exhaled air; Heated tobacco products
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Randomised controlled cross-over study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heated tobacco product (Experimental): 30 puffs of heated tobacco product IQOS
  Interventions: Other: Heated tobacco product
- Sham (Experimental): sham heated tobacco product
  Interventions: Other: Heated tobacco product

INTERVENTIONS:
Other: Heated tobacco product — Sham heated tobacco product

SUMMARY:
This is a human randomized controlled cross-over study where we investigate the effects of heated tobacco products (HTP) on lung function and on assessing volatile organic compounds in exhaled air.

DETAILED DESCRIPTION:
The World Health Organization estimates that smoking is one of the leading causes of premature death worldwide with an estimated 5-8 million lives lost annually due to tobacco usage.

Heated tobacco products (HTP) is a new form of tobacco products. HTP usually consists of a pod with tobacco that is mixed with glycerol which is inserted into a heating chamber. HTP is not combusted but only heated. Previous studies into smoking cessation with regular cigarettes and electronic cigarettes have suggested a risk for double usage instead of cessation, augmenting a nicotine addiction. There is a risk that HTP use simply enhances nicotine usage and smoking addiction.

There is limited data on the health effects of HTP. A majority of the studies available have reported conflicts of interest to manufacturers of HTP. It has been shown that aerosols from HTP contain toxic compounds and free radicals just as in regular cigarette smoke, albeit in lower concentrations (6-8). Furthermore, aerosols from HTP can spread in a room, enabling passive exposure (9). It has been shown that there is a decrease in harmful biomarkers in smokers that switch to HTP after 5 days of usage but also of a higher HTP consumption compared to regular smoking. There are few studies on effects of HTP in humans. We seek to assess the effects of HTP usage on lung function and the presence of volatile organic compounds in exhaled air using non invasive methods.

Subjects and criteria:

Twenty five male or female occasional tobacco users (age 18-40, maximum 10 cigarettes per month or 10 pouches of snus per month) will be included. They have to be healthy, having no preexisting conditions or take any medications. All subjects will have to complete a normal health declaration.

Methods:

In randomized cross-over fashion subjects will either inhale vapor (1 puff per minute for 30 minutes, total 30 puffs) from a HTP of the brand IQOS (IQOS 3 Multi, Philip Morris AB) or perform sham-smoking of HTP.

Baseline coitinine in the blood and volatile organic compounds in exhaled air will be measured. Subjects will then use HTP as described above. Exhaled air is collected following exhaling a full breath by the volunteer at normal speed through a disposable mouthpiece connected to an open 129 ml plastic cylinder with valve and manual piston (Bio-VOC-2 breath sampler, Markes International). The valve has a low resistance which makes it very easy to blow air through the cylinder. A filter cassette with gas sampling tubes is then connected to the cylinder where the last 129 ml of the exhaled air remains. Using the piston, the air is then emptied onto the pipe via the filter. The gas sampling tube and the filter are marked with unique markings, which can then be linked to a sample code. The procedure can now be repeated 1-4 times to collect additional exhaled air. The total sampling time is from 2-7 minutes depending on the number of repetitions. After each exposure, exhaled air is collected 3-4 times for approximately two hours.

The gas sampling tube contains an inert adsorbent material which, when heated (~ 300 ° C) in a oxygen-free carrier gas, releases the volatile organic substances trapped during sampling. The substances are then analyzed using gas chromatography connected to a mass spectrometer, where the intensity of the substances' different mass / charge ratios is collected. After calibrating the instrument's response to various substances, the concentration in the exhaled air is calculated. For substances where there is no reference substance, a quantification is performed against a reference substance with a known response factor and identification is carried out with criterion requirements for match factor by means of a deconvolution program (AMDIS) against data in a mass spectrum reference library from NIST. Preliminary own tests and method comparisons with previous studies indicate that the data material will contain in the order of 30-100 identified volatile organic compounds.

Specification of VOCs:

The exhaled air is analyzed for the following VOCs:

Acetaldehyde Acetic acid Acetic acid, methyl ester Acetone Acetonitrile Acetophenone Acrolein alpha-Pinene Benzaldehyde Benzene Benzene, 1-chloro-4-methyl- Benzene, bromopentafluoro- Benzoic acid Benzonitrile Butanal Butane, 2,3-dimethyl-2,3-dinitro- Butanoic acid, methyl ester Cyclohexane Cymene Decanal Decane Diethyl carbitol D-Limonene Etanol Ethene, 1,1-dichloro- Ethylbenzene Formamide, N,N-diethyl- Furan, 2-methyl- Furan, tetrahydro-3-methyl- Heptanal Hexanal Hexane Hexane, 2,2-dimethyl- Hexane, 3-methyl- Hexanoic acid Isoprene Isopropyl Alcohol Methacrolein Methanol Methylene chloride N-Ethylformamide Nitrogen gas Nonanal Nonane Octanal Octane p-Cymene Phenol Phthalic anhydride Propane, 1-(methylthio)- p-Xylene Silane, triethylfluoro- Styrene Sulfide, allyl methyl Sulfur dioxide Tetrahydrofuran Toluene Triethyl phosphate Undecanal 1,3-Dioxolane, 2-methyl-

1-Dodecene

1. H-Pyrrole, 1-ethyl- 1-Propene, 1-(methylthio)-, (E)- 1-Propene, 2-methyl- 2,2-Dimethoxybutane 2,3-Butanedione 2-Butanone 2-Ethylacrolein 2-Pentanone 2-Propanol, 2-methyl- 3-Pentanone 5-Hepten-2-one, 6-methyl-

ELIGIBILITY:
Inclusion Criteria:

• Healthy, free from medication

Exclusion Criteria:

* Any form of cardiovascular disease
* Any form of pulmonary disease like asthma or COPD
* Any form of systemic or chronic disorder like rheumatologic or metabolic diseases. - Symptoms of infection or inflammation within 4 weeks of the study
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Volatile organic compounds in exhaled air, nanogram/l (please see study description for specification of VOC) | preexposure
  in exhaled air
Volatile organic compounds in exhaled air, nanogram/l (please see study description for specification of VOC) | 10 minutes
  in exhaled air
Volatile organic compounds in exhaled air, nanogram/l (please see study description for specification of VOC) | 30 minutes
  in exhaled air
Volatile organic compounds in exhaled air, nanogram/l (please see study description for specification of VOC) | 120 minutes
  in exhaled air

CONTACTS AND LOCATIONS:
Locations (1):
- Institutionen för kliniska vetenskaper, Danderyds sjukhus, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No